CLINICAL TRIAL: NCT03843450
Title: Culture System for Isolating Circulating Tumor Cells
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201811053RINA
Record Dates: First submitted 2019-02-14; First posted 2019-02-18 (Actual); Last update posted 2020-11-05 (Actual); Status verified 2020-09

CONDITIONS: Early Detection of Cancer
Keywords: circulating tumor cells,WBCs adhesion, biomedical materials

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This culture system utilizes the special affinity difference of biomedical material coating for different cells to achieve the effect of isolating cancer cells from the blood sample. The coating of the system has the characteristic that to make the WBCs adhesion, but the cancer cells in the blood sample suspend in the culture medium, which achieves the effect of separating cancer cells from the blood. The supernatant with the cancer cells can further be isolated from the cultural system for related analysis and detection to achieve early diagnosis and screening.

ELIGIBILITY:
Inclusion Criteria:

1. Polycythemia patients are between the ages of 20 and 70.
2. Willing to sign the consent form under the informed consent.

Inclusion Criteria:

Exclusion Criteria:

1. Vulnerable Subjects included minors, prisoners, aborigines, pregnant women, people with mental disorders, students, and subordinates, etc.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include polycythemia patients between the ages of 20 and 70. We just use the waste blood from patients' routine phlebotomy therapy. Also, to protect the vulnerable subjects, we don't recruit minors, prisoners, aborigines, pregnant women, people with mental disorders, students, and subordinates, etc.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2019-01-29 (Actual); Primary Completion 2022-07-01 (Estimated); Study Completion 2022-09-26 (Estimated)

PRIMARY OUTCOMES:
Cancer Cell Isolation Efficiency of The Isolation System | 1 day
  The percentage isolation of fluorescently-labeled A549 cell lines will be spiked into the whole blood, and the put into the system. The supernatant of the system will be collected to re-culture on the culture dishes and analyzed by fluorescence microscope.
WBCs adhesion ratio | 1 hour
  The whole blood will be diluted and put into the system. And the supernatant will be collected to count the number of blood cell number by the automatic blood cell count.

CONTACTS AND LOCATIONS:
Overall Officials: Tai-Horng Young, Principal Investigator — Institute of Biomedical Engineering, National Taiwan University
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan